CLINICAL TRIAL: NCT01521572
Title: Effect of the Use of Salbutamol on the Mechanical Properties of the Respiratory System of Healthy Individuals, Smokers and COPD Patients
Brief Title: Effect of the Salbutamol on Mechanical Properties of Respiratory System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Gerusa Maritimo da Costa, Master, Rio de Janeiro State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2927/2011; CEP2927/2011HUPE (Other: Ethics Committee in Research of HUPE)
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Smoking; Airway Obstruction
Keywords: chronic obstructive pulmonary disease,; bronchial reversibility,; bronchodilator,; respiratory impedance,; forced oscillation technique,; plethysmography,; spirometry; Diagnostic Techniques, Respiratory System
MeSH Terms: conditions — Smoking; Airway Obstruction; Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Salbutamol (Experimental): Short-acting bronchodilator for use in humans released by the Ministry of Health, widely used worldwide for the treatment of chronic obstructive pulmonary disease.
  Interventions: Drug: Salbutamol sulphate

INTERVENTIONS:
Drug: Salbutamol sulphate — bronchodilator test, beta2-agonist, short-acting, six hours duration, 400 micrograms.
  Other Names: Aerogold; GO/DRUGS/341/L; LOTE: YR1070

SUMMARY:
The aim of this study is to assess the bronchodilator response of salbutamol on respiratory mechanics of healthy individuals, smokers and COPD with varying degrees of airway obstruction.

DETAILED DESCRIPTION:
Clinical evaluation will be conducted and anthropometric measurements, then the pulmonary function tests: forced oscillation technique (FOT), whole body plethysmography, spirometry and-administration of salbutamol aerosol for assessment of bronchodilator response. After 20 minutes, the individual will be evaluated again following the same sequence.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals, smokers and patients with chronic obstructive pulmonary disease.

Exclusion Criteria:

* healthy subjects: no history of smoking respiratory infection and disease respiratory
* smokers and chronic obstructive pulmonary disease patients: asthma and other respiratory diseases.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-01 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory function test | two o'clock
  Evaluation of pulmonary mechanics before and after salbutamol (short-acting bronchodilator) in healthy individuals, smokers and chronic obstructive pulmonary disease in stages: mild, moderate, severe and very severe according to GOLD criteria.

SECONDARY OUTCOMES:
Salbutamol | twenty minutes
  In the bronchodilator test will be used 400 micrograms of beta2-agonist short-acting. They will be asked to exhale slowly until they can no longer expel more air from the lungs. To place the inhaler with a spacer between the lips, pressing them well, but no bite. Shortly thereafter start to breathe through the mouth and will be released a jet of 100 micrograms of the bronchodilator. Then they will hold their breath for 10 seconds. 3 puffs are made with 1 minute interval between each application.

CONTACTS AND LOCATIONS:
Overall Officials: Gerusa M Costa, MSc, Principal Investigator — State University of Rio de Janeiro; Pedro L Melo, PhD, Study Director — Laboratory biomedical instrumentation
Locations (1):
- Laboratory biomedical instrumentation - State University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- See also: http://www.ncbi.nlm.nih.gov/pubmed?term=gerusa%20maritimo%20da%20costa — http://www.ncbi.nlm.nih.gov